CLINICAL TRIAL: NCT07033429
Title: The Impact of Thiol-Disulfide Homeostasis and Ischemia-Modified Albumin Levels on In Vitro Fertilization Outcomes in Couples With Male Factor Infertility
Brief Title: Effect of Thiol-Disulfide Homeostasis and Ischemia-Modified Albumin Levels on IVF Results in Male Factor Infertility
Acronym: IVF
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Ali Yavuzcan, M.D., Professor, Duzce University
Other Study IDs: E-23-3605
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2023-04

CONDITIONS: The Serum Native Thiol (NT); Total Thiol (TT); Serum Disulfide/TT Ratio; NT/TT Ratio; Serum Ischemia-modified Albumin (IMA)
Keywords: infertility; in vitro fertilization; ischemia-modified albumin; male factor; thiol-disulfide homeostasis; unexplained
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Serum samples were collected from the males on the day of oocyte pick-up. Blood samples were drawn from the antecubital vein and transferred into gel-based biochemistry tubes for the determination of TDH, IMA and other biochemical parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: undergoing IVF due to male factor infertility
- control group: undergoing IVF due to unexplained infertility

SUMMARY:
Thiol-disulfide Homeostasis (TDH) is essential for physiological functions in the human reproductive system, including antioxidant defense, detoxification, signal transduction, enzymatic regulation, apoptosis, and cellular communication. Ischemia-Modified Albumin (IMA) serves as an indicator of oxidative stress (OS) and is linked to ischemia-reperfusion injury. This study aimed to investigate changes in OS markers, particularly TDH and IMA levels, in couples with male infertility, and to examine the relationship between these markers and in vitro fertilization (IVF) success. Understanding how TDH and IMA levels influence IVF outcomes is crucial for advancing reproductive treatments for couples having diagnosis of infertility.

DETAILED DESCRIPTION:
The thiol-disulfide Homeostasis (TDH) is believed to participate in critical physiological functions, including antioxidant defense, detoxification, signal transduction, enzymatic activity regulation, apoptosis, and cellular communication within the human reproductive system. Ischemia-Modified Albumin (IMA) is considered a surrogate marker for oxidative stress (OS) and has also been linked to ischemia-reperfusion injury. The present study was designed to investigate the alteration of OS markers, including TDH and IMA levels, in couples diagnosed with male infertility, and to examine the association between these OS markers and in vitro fertilization (IVF) success. Couples in which women aged 23-45 years and undergoing IVF treatment due to male factor and unexplained infertility will be enrolled. The serum native thiol (NT), total thiol (TT) levels, disulfide levels and disulfide/TT and NT/TT ratios will be compered between two groups. The serum ischemia-modified albumin (IMA) level will also compared between male infertility and unexplained infetility group. TDH related parameters as NT and TT may be useful as a reflection of OS and as potential diagnostic biomarkers for male infertility

ELIGIBILITY:
Inclusion Criteria: Couples in which women aged 23-45 years and undergoing IVF treatment due to male factor and unexplained infertility were enrolled.

-

Exclusion Criteria: Patients with hepatic or renal disease, systemic infections, systemic inflammatory disorders (such as diabetes mellitus, thyroid hormone disorders, rheumatologic, autoimmune, endocrine, neoplastic or other inflammatory conditions), or a diagnosis of endometriosis were excluded from the study. Smokers were excluded. Additionally, women with diminished ovarian reserve (DOR) were also not included in this study.

-

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples in which women aged 23-45 years and undergoing IVF treatment due to male factor and unexplained infertility were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Live birth rate (LBR) | 6 months
  live births to the total number of embryo transfer cycles
beta-human chorionic gonadotropin (hCG) positivity | 6 months
  serum ≥ 10 mlU/mL
clinical pregnancy (CP) | 6 months
  the detection of a gestational sac via transvaginal ultrasonography

SECONDARY OUTCOMES:
diagnosing male infertility | 6 months
  The serum native thiol (NT) levels, serum total thiol (TT) levels in males

CONTACTS AND LOCATIONS:
Overall Officials: Müzeyyen Gülnur Özakşit, M.D., Professor, Study Director — Ankara Bilkent City Hospital, IVF Unit
Locations (1):
- Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All of the data including demographic characteristics and laboratory findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the beginning of study up to now.

REFERENCES:
- [Background] Micoogullari U, Cakici MC, Kilic FU, Kisa E, Ozcift B, Caglayan A, Neselioglu S, Karatas OF, Erel O. Evaluation of the role of thiol / disulfide homeostasis in the etiology of idiopathic male infertility with a novel and automated assay. Syst Biol Reprod Med. 2022 Apr;68(2):162-168. doi: 10.1080/19396368.2021.2003481. Epub 2021 Dec 10. PMID 34893004
- [Background] Zec I, Goldstajn MS, Kuna K, Mikus M, Stabile G, Bianco B, Buzzaccarini G, Lagana AS. Oxidative homeostasis in follicular fluid and reproductive outcomes - from bench to bedside. Prz Menopauzalny. 2022 Dec;21(4):276-284. doi: 10.5114/pm.2022.124019. Epub 2022 Dec 30. PMID 36704764
- [Background] Ozdemir AZ, Karli P, Neseli Oglu S. Does thiol/disulfide homeostasis affect the number of metaphase 2 oocyte in the treatment of in vitro fertilization? Future Sci OA. 2020 Jan 14;6(2):FSO452. doi: 10.2144/fsoa-2019-0132. PMID 32025332